CLINICAL TRIAL: NCT00596115
Title: Open Label Extension for Treating ALS With R(+) Pramipexole at 60 Milligrams Per Day
Brief Title: Treating Amyotrophic Lateral Sclerosis (ALS) With R(+) Pramipexole Dihydrochloride Monohydrate at 60 mg/Day
Status: Temporarily not available | Type: Expanded Access
Sponsor: Bennett, James P., Jr., M.D., Ph.D. (Individual)
Collaborators: University of Pittsburgh (Other); University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 12316
Record Dates: First submitted 2008-01-05; First posted 2008-01-16 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

INTERVENTIONS:
Drug: R(+) pramipexole dihydrochloride monohydrate — 20 mg tid per day orally

SUMMARY:
R(+) pramipexole dihydrochloride monohydrate [R(+)PPX], an experimental neuroprotective drug, is provided in this open label extension study to ALS patients who have participated in earlier clinical protocols.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of ALS

Exclusion Criteria:

* No prior participation in R(+)PPX clinical studies

Ages: 30 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult